CLINICAL TRIAL: NCT07007715
Title: Optimizing High-flow Nasal Cannula Settings: Comparing Different Flow Approaches and Exploring Physiological Phenotyping With End-expiratory Lung Volume, Peak Tidal Inspiratory Flow and Oxygen Demand
Brief Title: Identifying the Best Flow Setting Strategy for High-Flow Nasal Cannula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Sheng-Yuan Ruan, MD, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202502078RINA
Record Dates: First submitted 2025-05-18; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Extubation Readiness; Respiratory Failure With Hypoxia
Keywords: flow rate; high flow nasal cannula; peak inspiratory flow; reintubation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Flow of 40L/min (Active Comparator): Setting HFNC flow at 40 L/min
  Interventions: Other: Flow of 40L/min
- Peak tidal inspiratory flow (PTIF) guided (Experimental): Setting HFNC flow at 5 L/min above the peak tidal inspiratory flow (PTIF), up to a maximum of 60 L/min.
  Interventions: Other: Peak tidal inspiratory flow (PTIF) guided
- PaO2/FiO2 ratio guided (Experimental): Setting HFNC flow according to P/F ratio prior to extubation. Flow will be set at 60, 50 40 L/min if P/F ratio <250 mmHg, 250-300 mmHg and >300 mmHg, respectively.
  Interventions: Other: PaO2/FiO2 ratio guided
- Flow of 60L/min (Experimental): Setting HFNC flow at 60 L/min
  Interventions: Other: Flow of 60L/min

INTERVENTIONS:
Other: Flow of 40L/min — Setting flow rate at 40L/min
  Arms: Flow of 40L/min
Other: Peak tidal inspiratory flow (PTIF) guided — Setting HFNC flow at 5 L/min above the peak tidal inspiratory flow (PTIF), up to a maximum of 60 L/min.
  Arms: Peak tidal inspiratory flow (PTIF) guided
Other: PaO2/FiO2 ratio guided — Setting HFNC flow according to P/F ratio prior to extubation. Flow will be set at 60, 50 40 L/min if P/F ratio <250 mmHg, 250-300 mmHg and >300 mmHg, respectively.
  Arms: PaO2/FiO2 ratio guided
Other: Flow of 60L/min — Setting flow rate at 60L/min
  Arms: Flow of 60L/min

SUMMARY:
The goal of this randomized trial is to compare four different flow-setting approaches for post-extubation use of high-flow nasal cannula (HFNC). Selecting the appropriate flow rate when initiating HFNC oxygen therapy is both crucial and challenging for clinicians, as the physiological benefits of HFNC depend significantly on the flow rate. To date, there are no guidelines or consensus on flow-rate setting and weaning for HFNC oxygen therapy.

The investigators hypothesized that physiological marker-guided flow setting using peak tidal inspiratory flow (PTIF) or PaO₂/FiO₂ ratios lead to better extubation outcomes as compared to empirical flow setting of 40 L/min or 60 L/min.

Participants will be randomly assigned to one of four study groups with different flow setting strategies summarized as follows: (1) Setting flow at 40 L/min, (2) Setting flow at 5 L/min above the peak tidal inspiratory flow, up to a maximum of 60 L/min. (3) Setting flow according to P/F ratio prior to extubation. Flow will be set at 60, 50 40 L/min if P/F ratio <250 mmHg, 250-300 mmHg and >300 mmHg, respectively. (4) Setting flow at 60 L/min.

DETAILED DESCRIPTION:
High-flow nasal cannula (HFNC) is a promising intervention for post-extubation oxygen therapy, with the potential to improve oxygenation, increase end-expiratory lung volume (EELV), reduce the work of breathing, and lower the risk of reintubation. Selecting an appropriate flow rate when initiating HFNC therapy is both crucial and challenging for clinicians. Although the physiological benefits of HFNC depend significantly on the flow rate, arbitrarily applying higher flow rates without appropriate patient selection may increase the risk of barotrauma and patient discomfort. Currently, there are no established guidelines or consensus on flow-rate setting for HFNC therapy. Given the growing use of HFNC, determining the optimal flow-setting strategy is urgently needed to ensure both clinical efficacy and cost-effectiveness.

This 4-arm parallel-group randomized trial aims to compare four different flow-setting approaches for post-extubation use of HFNC in extubation outcomes. The individual flow-setting strategy for each study arm is summarized as follows: (1) Setting flow at 40 L/min, (2) Setting flow at 5 L/min above the peak tidal inspiratory flow, up to a maximum of 60 L/min. (3) Setting flow according to P/F ratio prior to extubation. Flow will be set at 60, 50 40 L/min if P/F ratio <250 mmHg, 250-300 mmHg and >300 mmHg, respectively. (4) Setting flow at 60 L/min. In addition, this study will incorporate measurements of peak tidal inspiratory flow and EELV to highlight the physiological characteristics of individual patients. These physiological measures may serve as both explanatory variables and potential predictors of flow responders. By examining the associations among flow responders, peak tidal inspiratory flow, pre-extubation oxygen demand, and changes in EELV, we aim to develop a comprehensive understanding of the mechanisms and key factors influencing flow responsiveness during post-extubation care with HFNC.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and receiving mechanical ventilation for more than 24 hours
* Ready for planned extubation after passing a spontaneous breathing trial
* PaO2/FiO2 <350 mmHg on the day of extubation

Exclusion Criteria:

* Age <18 years
* On do-not-reintubate code
* Pregnant women
* Having tracheostomies
* Infeasibility of using HFNC
* Planning to use preventive NIV after extubation by the primary care team
* Life expectancy less than one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
A composite outcome of noninvasive ventilation (NIV) use or reintubation within five days after extubation | 5 days
  A single global test of significance to compare between-group difference in the composite outcome

SECONDARY OUTCOMES:
Proportion of reintubation within five days after extubation | 5 days
  A single global test of significance to compare between-group difference in proportion of reintubation within five days
Proportion of NIV use within five days after extubation | 5 days
  A single global test of significance to compare between-group difference in proportion of NIV use within five days.
28-day mortality | 28 days
  28-day mortality
Change in PaO2/FiO2 ratio between 0 and 24th hour | 24 hours
  Change in PaO2/FiO2 ratio between 0 and 24th hour
Change in arterial CO2 level (mmHg) between 0 and 24th hour | 24 hours
  Change in arterial CO2 level (mmHg) between 0 and 24th hour
Proportion of ahead-of-schedule change in flow rates in 24 hours | 24 hours
  Proportion of ahead-of-schedule change in flow rates in 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided